CLINICAL TRIAL: NCT07115524
Title: Comparative Accuracy of Activity Scores of Intestinal Ultrasound and Colonoscopy in Monitoring Ulcerative Colitis Activity
Acronym: IUS/IBD
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Mohammed Abdel Mowgod, Lecturer in Tropical Medicine and Gastroenterology, Assiut University
Other Study IDs: 4-2025-300644
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-08

CONDITIONS: AssessIUS Scores inUC Versus Colonoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our study aimed to assess simple sonographic activity scores and Colonoscopy for active UC patients

DETAILED DESCRIPTION:
Ulcerative colitis (UC) has a relapsing-remitting course which necessitates frequent follow-up examinations to monitor disease activity.

Disease management was previously guided by patient reported symptoms, and treatment targets were based on symptom control. However, the patient's symptoms do not necessarily correspond to inflammatory activity and current guidelines recommend that management should be based on objective evaluations.

Ileocolonoscopy is considered the reference standard method for determining disease status in Ulcerative colitis. Although validated and reproducible scoring systems are complex and cumbersome to use in clinical practice, and even though ileocolonoscopy is an excellent tool for activity monitoring, it cannot be performed on a regular basis as it is invasive, is resourceintensive and causes considerable patient discomfort. As numerous follow-up examinations are required, simple non-invasive surrogate markers are needed.

Biomarkers such as C-reactive protein [CRP] and faecal calprotectin are well established in both primary work-up and disease monitoring.

Still, as they cannot depict disease location and have limited accuracy, additional tools are required.

Gastrointestinal ultrasound [GIUS] has high diagnostic accuracy for detecting active CD, and in trained hands, it can make significant impact on clinical decision-making.

Furthermore, as it is non-invasive, readily available and can be performed bedside, the modality seems well suited for bedside and frequent activity monitoring.

Still, interpretation of the GIUS findings may be influenced by the sonographer's level of experience. A standardized ultrasound activity index may simplify the interpretation of the sonographic findings, allowing for easier comparison between different examinations during follow-up. Although various sonographic activity scores are available, the methodology for development was shown to be insufficient in most studies and no index is in widespread clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Any patient above age of 18 years old and diagnosed to have active UC through:
* Clinical features: rectal bleeding, with frequent stools and mucous discharge from the rectum. Some patients also describe tenesmus. The onset is typically insidious.
* Endoscopic findings include the following; loss of vascular pattern, Granular and fragile mucosa, friability, ulcerations, erosions, pseudo-polyposis

Exclusion Criteria:

* Patients with UC who are under age of 18 years' old.
* Pregnancy.
* Previous colectomy.
* Patient refuse to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: -Thorough medical history including abdominal pain, bloody diarrhea and its frequency, tensesmus,and mucous with stool, and physical examination (general and abdominal) stressing on fever, tachycardia, abdominal tenderness and significant weight loss. Each patient was phenotypically classified according to the Montreal classification (14).
  Harvey Bradshaw Index [HBI] (15) was used to assess clinical disease activity, where clinical remission was defined as HBI < 5.
  * Colonoscopy will done and assessment of severity according to Mayo Endoscopic Score (MES) for ulcerative colitis.
  * Intestinal ultrasound examination:
  * Patient preparation: no specific preparation needed but fasting 6-8 hours before examination decrease gaseous content and allow better visualization.
  * Calculate ultrasound activity scores (including Ulcerative Colitis-Intestinal Ultrasound Index (UC-IUS index), Simple IUS score).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Correlation Between Simple Sonographic Activity Scores and Colonoscopy Findings in Active Ulcerative Colitis | At baseline (Day 0) from hospital admission
  To evaluate the relationship between intestinal ultrasound (IUS)-based sonographic activity scores and endoscopic disease activity assessed by colonoscopy in patients with active ulcerative colitis. The aim is to determine whether sonographic scoring can serve as a non-invasive surrogate for endoscopic assessment in monitoring disease activity.
Assessment of Sonographic Activity Scores Compared to Colonoscopy in Active Ulcerative Colitis Patients | At baseline (Day 0 of hospital admission)
  To evaluate the diagnostic accuracy and clinical relevance of simple intestinal ultrasound (IUS) activity scores in assessing disease activity in patients with active ulcerative colitis (UC), using colonoscopy findings as the reference standard.